CLINICAL TRIAL: NCT00152906
Title: Phase I/II Trial of Highly Conformal Radiotherapy for Unresectable Liver Metastases and Hepatobiliary Carcinoma
Brief Title: Stereotactic Radiotherapy (SRT) Liver (COLD 1)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: American Society of Clinical Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 03-0295-C; ASCO Clinical Research Grant
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Liver Neoplasms; Neoplasm Metastases
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis | interventions — Radiosurgery

ARMS (1):
- Stereotactic RT or highly conformal RT (Experimental)
  Interventions: Procedure: Stereotactic radiotherapy (SRT) or highly conformal (CRT)

INTERVENTIONS:
Procedure: Stereotactic radiotherapy (SRT) or highly conformal (CRT) — SRT or CRT is radiation delivered precisely conforming the high dose region to the tumor, usually in a few highdose fractions.

SUMMARY:
A minority of patients with colorectal liver metastases and hepatobiliary cancer (primary liver cancer) are candidates for surgery, but there are no curative treatment options for these patients. Their median survival time is 3 to 12 months. Stereotactic radiation (SRT) (highly conformal radiotherapy (CRT)) is a treatment option for these patients with unresectable liver cancer, now possible due to improvements in our ability to localize and immobilize liver tumors and an improved understanding of the partial liver volume tolerance to radiation. SRT should permit liver tumors to be treated to tumorcidal doses while sparing the uninvolved liver, decreasing the risk of treatment related normal tissue toxicity. With such conformal radiation, it is possible to deliver radiation in fewer fractions than traditionally required, which should be more convenient for patients. In this study, CRT will be delivered during shallow breathing or breath hold to minimize organ motion due to breathing, decreasing the volume of normal liver that must be irradiated.

ELIGIBILITY:
Inclusion Criteria:

* Primary hepatobiliary confirmed pathologically or via imaging
* Liver metastases from colorectal cancer or other solid malignancy, confirmed pathologically
* New radiographic liver lesions most consistent with metastases, in a patient with previously pathologically proven solid malignancy and a previously negative liver contrast CT or MRI
* The tumor must be unresectable or the patient must be medically inoperable or extra-hepatic metastases must be present
* Karnofsky performance status (KPS) > 60
* Age > 18 years
* Patients must have recovered from the effects of previous surgery, radiotherapy or chemotherapy
* Chemotherapy must be completed at least 2 weeks prior to radiation therapy or not planned to be administered for at least 2 weeks
* Adequate organ function as assessed as follows:Hemoglobin > 90 g/L, Absolute neutrophil count > 1.5 bil/L, Platelets > 80,000 bil/L, Bilirubin < 3.0 times upper range of normal, INR < 1.3 or correctable with vitamin K, AST or ALT < 6.0 times upper range of normal, Creatinine < 200 umol/L (other than patients who are having dialysis or already have dialysis lines in place for future dialysis for renal failure. These patients may be treated on study with no upper limit on their creatinine.)
* Child A liver score
* Previous liver resection or ablative therapy is permitted.
* Life expectancy > 3 months
* Multiple metastases are permitted (volume of uninvolved must be at least 800 cc, and the maximal effective liver volume that may be treated is 80%.
* Informed consent form

Exclusion Criteria:

* Patients with active hepatitis or clinically significant liver failure
* Prior radiation therapy to the right upper abdomen, precluding re-irradiation of the liver. (Prior pelvic radiation is permitted, as long as no overlap between pelvic and liver radiation fields occurs.)
* Prior uncontrolled, life threatening malignancy within the past year.
* Gross (clinically apparent) ascites.
* Pregnancy is not permitted, and in women of child bearing age, a pregnancy test and birth control are warranted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2003-07; Primary Completion 2016-07 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Phase I: To evaluate feasibility and maximally tolerated dose of SRT | assessment: weekly during treatment; 1, 3, 6, 9, 12 months post, every 6 months for up to 3 years
Phase II: To determine with more confidence the rate and spectrum of all toxicities that occur at the maximally tolerated dose of radiation. | assessment: weekly during treatment; 1, 3, 6, 9, 12 months post, every 6 months for up to 3 years

SECONDARY OUTCOMES:
To evaluate local control, progression-free survival and survival of patients with unresectable primary hepatobiliary cancer and metastatic liver cancer treated with SRT. | assessment: weekly during treatment; 1, 3, 6, 9, 12 months post, every 6 months for up to 3 years
To evaluate the quality of life. | assessment: pre-treatement, 1, 3, 6,12 months post
To evaluate changes in liver function following SRT. | 3 to 12 months
To evaluate patterns of breathing at and during RT. | during radiation treatment only
To develop more confidence in a revised normal tissue complication probability (NTCP) model for radiation induced liver toxicity and collect preliminary data to determine how the liver responds to radiation. | at 3 months post RT
To determine whether serum cytokines and P-III-P can help predict RILD. | baseline, during radiation and up to 3 months post radiation

CONTACTS AND LOCATIONS:
Overall Officials: Laura Dawson, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Bujold A, Massey CA, Kim JJ, Brierley J, Cho C, Wong RK, Dinniwell RE, Kassam Z, Ringash J, Cummings B, Sykes J, Sherman M, Knox JJ, Dawson LA. Sequential phase I and II trials of stereotactic body radiotherapy for locally advanced hepatocellular carcinoma. J Clin Oncol. 2013 May 1;31(13):1631-9. doi: 10.1200/JCO.2012.44.1659. Epub 2013 Apr 1. PMID 23547075